CLINICAL TRIAL: NCT05845723
Title: Efficacy and Safety of Tocilizumab and Tofacitinib in the Treatment of Patients With Vascular Behçet's Syndrome
Brief Title: Tocilizumab and Tofacitinib in the Treatment of Vascular Behçet's Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCZ/TOF-VBS-PUMCH
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-07

CONDITIONS: Aneurysm; Behcet Syndrome, Vascular Type
Keywords: Tocilizumab; Tofacitinib; Vascular Behçet's Syndrome
MeSH Terms: conditions — Aneurysm; Behcet Syndrome | interventions — tocilizumab; tofacitinib; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tocilizumab+GCS for VBS (Experimental): Participants randomized to this arm will receive prednisone 1mg/kg/d, gradually tapered to 10mg/d at week 12, combined with intravenous infusion of tocilizumab 8mg/kg every 4 weeks for 24 weeks.
  Interventions: Drug: tocilizumab
- Tofacitinib+GCS for VBS (Experimental): Participants randomized to this arm will receive prednisone 1mg/kg/d, gradually tapered to 10mg/d at week 12, combined with oral tofacitinib 5mg twice a day for 24 weeks of treatment.
  Interventions: Drug: tofacitinib
- Cyclophosphamide+GCS for VBS (Experimental): Participants randomized to this arm will receive prednisone 1mg/kg/d, gradually tapered to 10mg/d at week 12, combined with intravenous infusion of cyclophosphamide 0.5g biweekly for 24 weeks.
  Interventions: Drug: cyclophosphamide

INTERVENTIONS:
Drug: tocilizumab — Participants will receive intravenous infusion of tocilizumab 8mg/kg every 4 weeks for 24 weeks.
  Other Names: ACTEMRA®
  Arms: Tocilizumab+GCS for VBS
Drug: tofacitinib — Participants will receive tofacitinib 5mg twice a day for 24 weeks of treatment.
  Other Names: Xeljanz®
  Arms: Tofacitinib+GCS for VBS
Drug: cyclophosphamide — Participants will receive intravenous infusion of cyclophosphamide 0.5g biweekly for 24 weeks.
  Other Names: Endoxana
  Arms: Cyclophosphamide+GCS for VBS

SUMMARY:
This project aims to evaluate the efficacy and safety of the combination of glucocorticoids with tocilizumab or tofacitinib, compared to the traditional combination of glucocorticoids with cyclophosphamide in the treatment of vascular Behçet's syndrome.

DETAILED DESCRIPTION:
Behçet's Syndrome (BS) is a recurrent and systemic vasculitis, with an incidence rate of about 14/100,000 in China, higher than that in Europe and America. Vascular Behcet's Syndrome (VBS) is an important subtype of BS characterized by multiple venous and artery lesions. It affects 20-25% of BS patients, predominantly young adult males, and is the leading cause of mortality in BS patients (67%), especially in patients with aneurysms. Therefore, exploring the diagnosis and treatment strategies for VBS is key to improving the prognosis of BS.

This project aims to investigate the efficacy and safety of the combination of glucocorticoids (GCS) with the biologic agent tocilizumab or the targeted small molecule tofacitinib, compared to the combination of GCS with cyclophosphamide in the treatment of VBS aneurysms, as well as to screen for biomarkers related to the response of tocilizumab or tofacitinib, and to improve the assessment and treatment of VBS and establish a precision diagnosis and treatment strategy.

This is a Phase IIb, multi-center, randomized, open-label, GCS plus cyclophosphamide-controlled, parallel design, prospective clinical study. Patients will be randomly assigned to three groups in a 1:1:1 ratio (tocilizumab + GCS vs tofacitinib + GCS vs cyclophosphamide + GCS, 27:27:27) after screening and recruitment. Patients will be followed up every 4 weeks from weeks 0-12, and every 6 weeks from weeks 12-24. The primary endpoint is the complete remission (CR) rate at the 12th-week follow-up. All participants will undergo their final visit at 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1． Understand and voluntarily sign an informed consent form prior to any study-related assessments/procedures being conducted.

2. Male and female subjects aged 18-65 years.

3． Fulfill the 2013 International Classification Criteria for Behcet's Disease (ICBD).

4． Patients with aneurysmal dilatation/aneurysm of the descending aorta and/or peripheral arteries confirmed by ultrasonography and/or computed tomography angiography (CTA).

5. Elevated acute phase reactants ESR and hs-CRP.

Exclusion Criteria:

1. Cardiovascular manifestations that cannot be distinguished from giant cell arteritis, Burger's disease, or atherosclerotic aneurysm; infectious aneurysm;
2. Other active organ involvement related to BS that requires intensified immunosuppressive treatment, including gastrointestinal ulcers, uveitis, and parenchymal neurological involvement;
3. Patients with severe aneurysms requiring emergency intervention surgery; patients with elective surgery indications require the consensus between rheumatologists and vascular surgeons to determine inclusion or exclusion.
4. Severe organ dysfunction, including ALT, AST, and TBIL exceeding the upper limit of normal by more than 2 times, serum creatinine ≥ 133 mmol/L, white blood cell count < 3×10^9/L, ANC < 2×10^9/L, hemoglobin < 80g/L, platelet count < 100×10^9/L;
5. Active infection such as active tuberculosis, hepatitis B or C, syphilis, chronic EBV infection, persistent or severe bacterial or viral infection;
6. Primary or secondary immunodeficiency;
7. Malignant tumor;
8. Use of immunosuppressants such as Cyclosporin A (CsA), Azathioprine (AZA), Tacrolimus (TAC), Mycophenolate Mofetil (MMF), or Cyclophosphamide (CTX) within 1 month;
9. Use of biologics/small molecule drugs within 5 half-lives (baricitinib within 10 days; etanercept within 4 weeks; infliximab within 8 weeks; adalimumab, golimumab, ustekinumab, and abatacept within 10 weeks, secukinumab within 6 months, and previously use of tocilizumab and tofacitinib);
10. Pregnant, lactating, or planning a recent pregnancy;
11. Subjects who do not agree to or are unable to comply with regular visits.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the complete response (CR) rate at week 12. | Baseline to week 12
  CR: the resolution of VBS-related symptoms and abnormal acute phase reactants including erythrocyte sedimentation rate (ESR) and high-sensitivity C reactive protein (hs-CRP), no progression or new occurrence of vascular lesions compared to baseline.

SECONDARY OUTCOMES:
The secondary endpoints include CR rate at week 24, and partial response (PR) rate at week 12/24. | Baseline to week 24
  PR: improvement in clinical symptoms, >50% decrease in inflammatory markers, no progression or new occurrence of vascular lesions.
Change From Baseline in Disease Activity as Measured by Behçet's Disease Current Activity Form (BDCAF). | BDCAF were assessed at weeks 0, 4, 8, 12, 18, and 24
  The BDCAF consists of 3 component scores: the Behçet's Disease Current Activity Index (BDCAI) score, the Patient's Perception of Disease Activity, and the Clinician's Overall Perception of Disease Activity. The BDCAI consists of 12 questions regarding disease manifestations over the previous 4 weeks, including oral and genital disease activity, as well as other manifestations of BS involving the skin, joints, GI tract, eyes, nervous system, and vascular system. The BDCAI score is the sum score of 12 items and ranges from 0 to 12. The Patient's Perception of Disease Activity and the Clinician's Overall Perception of Disease Activity were assessed on a scale from 1 to 7. A higher score indicates a higher level of disease activity (worsening), and a negative change from baseline indicates improvement.
Change From Baseline in the degree of vasculitis damage as Measured by Behçet's syndrome Overall Damage Index (BODI). | BODI were assessed at weeks 0 and 24
  The BODI consists of 4 overarching principles and 34 items with 12 subitems, categorized into 9 organ/system domains: mucocutaneous, musculoskeletal, ocular, vascular, cardiovascular, neuropsychiatric, gastrointestinal, reproductive system, and miscellaneous. Each item and subitem score 1 point. The total score ranges from 0 to 46. The higher the score, the greater the degree of damage.
4.Change From Baseline in the degree of vasculitis damage as Measured by Vasculitis Damage Index (VDI). | Time Frame: VDI were assessed at weeks 0, 12, and 24
  The VDI consists of 64 items, categorized into 11 organ/system domains: musculoskeletal, skin, ear, nose, and throat, pulmonary, cardiovascular, renal, gastrointestinal, peripheral vascular, ocular, neuropsychiatric, and other damage. Each item scores 1 point. The total score ranges from 0 to 64. The higher the score, the greater the degree of damage.
Change From Baseline in ESR and hs-CRP. | ESR and hs-CRP were assessed at weeks 0, 4, 8, 12, 18, and 24
  The ESR and hs-CRP are acute phase reactants that are indicative of the patient's degree of disease activity.
6.Change From Baseline in imaging changes including vascular ultrasonography, and CTA (including progression, improvement, and stability) | Imaging examinations were assessed at weeks 0, 12 and 24
  Radiological improvements is defined as the attenuation of radiological abnormalities related to VBS, including a reduction in aneurysm size. Radiological progression is defined as an increase in aneurysm size, aneurysm rupture, or the appearance of new lesions. Radiological stability is defined as the maintenance of aneurysm size and the absence of new lesions.
7.Change From Baseline in 36 health survey questionnaire (SF-36). | SF-36 were assessed at weeks 0, 12, and 24
  The SF-36 is primarily used to evaluate eight dimensions of health-related quality of life: physical functioning (PF), role limitations due to physical health problems (RP), bodily pain (BP), general health perceptions (GH), vitality (VT), social functioning (SF), role limitations due to emotional problems (RE), and mental health (MH). In addition, there is a health transition (HT) item that assesses the overall change in health status over the past year. SF-36 also includes another health indicator, Reported Health Transition, which is used to evaluate the overall change in health status over the past year. Higher scores indicate better health status.
Safety assessment: Record the types, frequency, and severity of adverse events, as well as the number of study participants who were discontinued due to any adverse events. | Adverse events were assessed at weeks 0, 4, 8, 12, 18, and 24
  Adverse event: Any medical condition that affects the health of the participant during the study or worsens a pre-existing medical condition, regardless of whether it is causally related to the study, is considered an adverse event. This can be symptoms, signs, or abnormal laboratory tests.
  Serious adverse event (SAE): Any significant medical event that causes death, is life-threatening, requires hospitalization, results in permanent or severe disability or loss of function, or the investigator deems it a significant medical event that may seriously harm the participant or require medical intervention to prevent the above outcomes. The causal relationship between the serious adverse event and the study is determined by the investigator's discussion.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No